CLINICAL TRIAL: NCT00341367
Title: Genetic Risk of Chronic Pain After Acute Sciatica
Brief Title: Blood Sample Donations to Study the Role of Genes in Pain
Status: Completed | Type: Observational
Sponsor: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999903070; 03-AA-N070
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-03-11

CONDITIONS: Pain
Keywords: Analgesic; Back Pain; Lumbar Disc; Nerve; Radiculopathy
MeSH Terms: conditions — Pain; Back Pain; Radiculopathy

SUMMARY:
This study attempts to identify genes that may increase or decrease the likelihood of sciatic pain (shooting pain down the leg) persisting 1 year after treatment of a herniated spinal disc. Many proteins in the nerves, spinal cord, and brain are involved in processing pain. These proteins vary slightly in different people. Animal studies have shown that rats and mice with certain types of proteins experience chronic pain after sciatic injury while those with other types do not. Better information about the role of genes in pain processing may lead to a test for the risk of chronic pain for specific individuals and more effective treatment approaches.

This study will include people who participated in the Maine Lumbar Pain Study of the natural history of spinal pain. The Maine study included patients treated for sciatic pain caused by a herniated disc. In this study, patients who did not improve with medical treatment were referred for surgery to remove the disc. Of those referred for surgery, 275 elected to have the operation, and 232 did not. One year after surgical consultation, leg pain was reduced in 81 percent of patients who underwent surgery. Of those who declined surgery, 56 percent improved after 1 year. This study will look for genetic differences in the non-surgical group that might reveal differences among those who improved and those who did not.

Participants will provide a blood sample (approximately 2 tablespoons) for genetic testing. They will also provide information on the ethnic background of their parents and grandparents. Different gene variants occur in different ethnic groups, so information on ethnic background will help researchers know what gene variants to look for. Participants will complete a questionnaire about their smoking history, because the same protein in the brain that responds to nicotine may also play a part in decreasing or increasing pain. Also, some surgeons believe that smoking can interfere with spinal bone healing. Information from this study will help resolve this question.

...

DETAILED DESCRIPTION:
Many patients have persistent pain one year after herniated lumbar disc even when the disc is surgically removed or shrinks spontaneously. We hypothesize that the risk of persistent pain is modified by common variations in genes related to inflammation and pain processing. We propose to collect blood for DNA analysis from up to 500 patients who have been followed for 10 years after the onset of severe sciatica in the Maine Lumbar Spine Study. Based on the pain research literature, Human Genome databases, and gene studies in NIAAA's Laboratory of Neurogenetics, we will prioritize approximately 100 candidate genes with variants that affect the function of their proteins. We will type patients' DNA for these variants and compare their clinical data with their genotype at each candidate gene to see if common variants increase or decrease the risk of chronic pain. The primary phenotype variable will be the amount of persistent leg pain one year after pain onset, Identification of such associations, if replicated in future studies, may help to prioritize targets for drug treatments or identify genetic tests that can predict the prognosis of acute sciatica and assist in treatment choice.

ELIGIBILITY:
* INCLUSION CRITERIA:

Presented to Maine orthopedic or neurosurgeon approximately 10 years ago with complaint of sciatica and was enrolled in Maine Lumbar Spine Study.

Outcome dataset includes ratings of low back and leg pain at baseline and at least one followup evaluation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2002-12-10; Study Completion 2010-03-11

CONTACTS AND LOCATIONS:
Locations (1):
- Maine Health Information Center, South Portland, Maine, United States

REFERENCES:
- [Background] Atlas SJ, Deyo RA, Keller RB, Chapin AM, Patrick DL, Long JM, Singer DE. The Maine Lumbar Spine Study, Part II. 1-year outcomes of surgical and nonsurgical management of sciatica. Spine (Phila Pa 1976). 1996 Aug 1;21(15):1777-86. doi: 10.1097/00007632-199608010-00011. PMID 8855462
- [Background] Atlas SJ, Keller RB, Chang Y, Deyo RA, Singer DE. Surgical and nonsurgical management of sciatica secondary to a lumbar disc herniation: five-year outcomes from the Maine Lumbar Spine Study. Spine (Phila Pa 1976). 2001 May 15;26(10):1179-87. doi: 10.1097/00007632-200105150-00017. PMID 11413434
- [Background] Deyo RA. Low-back pain. Sci Am. 1998 Aug;279(2):48-53. doi: 10.1038/scientificamerican0898-48. No abstract available. PMID 9674171